CLINICAL TRIAL: NCT02152176
Title: Titration Morphinique autocontrôlée Par le Patient Par un Dispositif mécanique à Usage Unique Versus Administration Par l'infirmière Chez Les Patients Ayant Une Douleur aiguë sévère Aux Urgences.
Brief Title: Morphine Titration by Patient Self-controlled by a Mechanical Device Versus Administration by the Nurse for Patients With Severe Acute Pain in the Emergency Department
Acronym: TACIDOU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOI 2013-08
Record Dates: First submitted 2014-05-22; First posted 2014-06-02 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Acute Pain
Keywords: pain; analgesia; morphine; PCA; Nurse
MeSH Terms: conditions — Acute Pain; Pain; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patient Controlled Analgesy group (Experimental): Titration of morphine by Patient Controlled Analgesy. The opioid titration will be performed by the patient using PCA (Vygon Freedom 5) according to the principle of self with a refractory period of 5 minutes.
  Interventions: Device: Titration of morphine by Patient Controlled Analgesy
- Control group (No Intervention): titration will be perform in the usual manner in accordance with the recommendations : a nurse will assess pain using a visual analog scale in the control group to assess the need for a new bolus of morphine

INTERVENTIONS:
Device: Titration of morphine by Patient Controlled Analgesy — PCA is never used for titration but only for relay of titration. Self-controlled analgesia by PCA is our intervention.
  Arms: Patient Controlled Analgesy group

SUMMARY:
Intense acute pain is a common reason for Emergency admittance and its management is one of the major public health goals.

In the recommendations formalized experts, it is recommended to use a protocol titration with morphine bolus of 2 mg (for patients less than 60 kg) or 3 mg (for patients over 60 kg) repeated every 5 minutes with a target of the Visual Analog Scale less than or equal to 30.

Despite these specific recommendations and a broad awareness of the teams, management of pain remains to be improved, the major difficulty of morphine titration at the emergency department being the availability of paramedical personnel to perform revaluations and reinjection. Thus, effective analgesia would be obtained in 50% of cases to 30 minutes.

The investigators want to study the self-controlled morphine titration by the patient by a mechanical device for single use (efficacy/safety).

ELIGIBILITY:
Inclusion Criteria:

* Admission to an emergency department
* Acute pain (Visual Analog Scale > 60)
* Able to assess pain using the numerical scale
* Prescription of morphine titration

Exclusion Criteria:

* Physical or mental disorders limiting the understanding and / or use of a PCA
* History of allergy to morphine / hypersensitivity to any component
* Long-term treatment morphine
* Opioid therapy administered prior to inclusion
* Analgesic treatment level 2 (codeine, tramadol, nefopam ...) administered prior to inclusion or planned
* History of Substance Abuse
* Severe respiratory insufficiency
* Severe hepatic impairment
* Head trauma
* Intracranial hypertension
* Uncontrolled epilepsy
* Pregnant or lactating
* Patient jailed
* Incapacitated adult under guardianship
* Incapable of giving informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale <30 | 30min
  Evaluate the effectiveness of the analgesia of morphine titration self-controlled by the patient using a PCA device for single use ("PCA" group) opposing to an opioid titration carried out by the nurse (group 'Control')

SECONDARY OUTCOMES:
Evaluate the effectiveness in the group Patient Controlled Analgesy | 4h
  * time to obtain effective analgesia from prescirption
  * consumption of morphine
  * Visual Analog Scale evolution
  * percentage of patients relieved defined by VAS <40, 1 hour after the prescription of opioid titration
Satisfaction | 4h
  * patient satisfaction
  * nurse satisfaction
  * time to prepare morphine titration

OTHER OUTCOMES:
Assess the safety in the group Patient Controlled Analgesy | 4h
  * adverse events du to morphine
  * adverse events du to medical/nursing support

CONTACTS AND LOCATIONS:
Overall Officials: ROY Pierre-Marie, MD-PhD, Study Chair — UH Angers; SCHOTTE Thibault, Physician, Principal Investigator — UH Angers
Locations (2):
- France (2):
  - SCHOTTE Thibault, Angers
  - CHOUKROUN Jacques, Le Mans